CLINICAL TRIAL: NCT02007161
Title: Supersaturation and Precipitation of Diclofenac in the Stomach of Healthy Volunteers
Acronym: DDD13DICLO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Jens Van Den Abeele, dhr., KU Leuven
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: EudraCT 2013-004636-29
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Supersaturation and Precipitation in the Stomach
MeSH Terms: interventions — Diclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutritional State (Active Comparator): Fed vs. Fasted State
  Diclofenac potassium 50 mg
  Interventions: Drug: Diclofenac potassium 50 mg
- Use of a PPI (Active Comparator): Nexiam (esomeprazole) 40 mg
  Diclofenac potassium 50 mg
  Interventions: Drug: Diclofenac potassium 50 mg

INTERVENTIONS:
Drug: Diclofenac potassium 50 mg — Diclofenac potassium 50 mg
  Other Names: Cataflam

SUMMARY:
Investigate the supersaturation and precipitation behaviour of diclofenac in the stomach of healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Age 20 - 35 years

Exclusion Criteria:

* Illness
* Acute / Chronic gastric disorder
* Use of medicine
* (possible) pregnancy
* Frequent exposure to X-rays during the past year
* HIV / Hepatitis B Virus or Hepatitis C Virus infection

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Area under the Concentration - Time Curve | Every 10 minutes for 2 h